CLINICAL TRIAL: NCT02421978
Title: Inflammation-Induced CNS Glutamate During Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Other Study IDs: IRB00080062; 1R21MH105897 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Cognitive dysfunction; Inflammation; Fatigue; Decreased motivation
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Inflammation; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytokine Multiplex, CRP, TRP, KYN, mRNA analysis, methylation analysis, and gene analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chemotherapy-treated breast cancer group: Female subjects with Stage I-III breast cancer treated with chemotherapy will complete the neuropsychiatric assessment battery, blood sampling, self-report forms and magnetic resonance spectroscopy (MRS) scans
- Non-Chemotherapy-treated breast cancer group: Non-chemotherapy treated female subjects with Stage I-III breast cancer will complete the neuropsychiatric assessment battery, blood sampling, self-report forms and magnetic resonance spectroscopy (MRS) scans
- Control group: Age and race-matched healthy women will complete the neuropsychiatric assessment battery, blood sampling, self-report forms and magnetic resonance spectroscopy (MRS) scans

SUMMARY:
The purpose of this study is to try and provide data linking the impact of increased inflammatory cytokines as a result of chemotherapy and their relationship with increased levels of CNS glutamate and related behavioral and cognitive consequences in breast cancer patients. The investigators will use neuropsychiatric assessments, blood sampling and Magnetic Resonance Spectroscopy (MRS) to collect study data.

DETAILED DESCRIPTION:
Approximately 70% of women with breast cancer experience behavioral and/or cognitive symptoms during treatment with chemotherapy and approximately 30% of women continue to experience these symptoms months to years after treatment completion. There is mounting data to suggest that inflammation may be involved and indicate that chemotherapy-treated breast cancer patients exhibit higher inflammatory markers than non-chemotherapy-treated patients, and inflammatory markers including interleukin (IL)-6 and soluble tumor necrosis factor (sTNFR2) have been associated with chemotherapy-induced depression and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients will have undergone surgery (lumpectomy or mastectomy) with or without neoadjuvant or adjuvant chemotherapy
* Age between 21-65 years

Exclusion Criteria:

* Taking trastuzumab

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients who are chemotherapy treated and non chemotherapy-treated and medically healthy women without breast cancer in the control group
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Ratio of Glutamate to Creatine | Baseline
  Single voxel MRS (Magnetic Resonance Spectroscopy) scans will be done to determine the glutamate levels in the dACC (dorsal anterior cingulate cortex), basal ganglia and hippocampus and the glutamate/ creatine (Glu/Cr) ratio will be calculated.MRS utilizes a magnetic field to look at magnetic nuclei, which absorb and re-emit electromagnetic energy in the presence of the magnetic field. By looking at the peaks in the resultant spectra the structure and concentration of metabolites can be determined.
Levels of peripheral blood markers of inflammation | Baseline
  Peripheral blood samples will be analyzed for levels of plasma c-reactive protein (CRP), tumor necrosis factor (TNF) and its soluble receptors (sTNFR1 and 2), interleukin (IL)-1 beta and the IL-1 receptor antagonist, and IL-6 and its soluble receptor (sIL-6R).
Cognitive dysfunction | Baseline
  Cognitive measures of processing speed, attention, executive function, memory and motivation will be assessed.
Behavioral assessments | Baseline
  Behavioral assessments will be done to assessed to measure depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia, United States